CLINICAL TRIAL: NCT03786666
Title: Vascular Ultrasound Evaluation of Atherosclerotic Plaques and the Success of Recanalization in Patients With Carotid Artery Stenosis and Occlusion
Brief Title: Ultrasound Evaluation of Carotid Artery Atherosclerotic Plaques and Recanalization
Status: Completed | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: The First Affiliated Hospital of Soochow University (Other); The First Hospital of Jilin University (Other); The First Affiliated Hospital of Shanxi Medical University (Other); The Second People's Hospital of Liaocheng (Unknown); Liaocheng Brains Hospital (Unknown); Lanzhou University Second Hospital (Other); First Hospital of China Medical University (Other); Dalian Municipal Central Hospital (Other); Peking University Third Hospital (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); Henan Provincial People's Hospital (Other); Shengli Oilfield Hospital (Other); Zhengzhou First People's Hospital (Unknown); Weihai Municipal Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: VUS-CAS
Record Dates: First submitted 2018-12-20; First posted 2018-12-26 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Stroke
Keywords: Stroke; Ischemia; Carotid artery Stenosis; CEA; Stenting; Ultrasound; Vulnerable plaque
MeSH Terms: conditions — Stroke; Ischemia; Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Carotid artery plaques removed by CEA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Carotid artery recanalization CEA or carotid artery stenting — Carotid artery recanalization CEA or carotid artery stenting

SUMMARY:
The purpose of this multiple-center study are: 1) To establish the ultrasound criteria for evaluating vulnerable plaques by comparing the plaque echo characteristics before CEA (carotid artery endarterectomy) and plaque specimen after CEA.

2) To establish the carotid artery recanalization strategies based on the evaluation results of carotid artery and intracranial artery by color doppler flow imaging and TCCS/TCD (transcranial color coded sonography/transcranial doppler).

3) To compare the success rate and the incidence of restenosis between CEA and carotid artery stenting.

DETAILED DESCRIPTION:
In this study, a total of 1000-1200 patients with carotid artery moderate (50-69%, with symptoms), severe (70-99%) stenosis (with or without symptoms) or occlusion who received either CEA or stenting are to recruited. Before carotid artery recanalization, CDFI (color duplex flow imaging) and TCCS/TCD are used to evaluate the structures and hemodynamic of carotid artery and intracranial artery. In addition, patients are to be followed up by ultrasound 1 week, 3 month, 6month and 1 year after recanalization.

1. Ultrasound examinations procedures: According to the guidelines of vascular ultrasonography published by the Stroke Prevention Engineering Committee, the National Health Commission of China in 2015. The plaque characteristics, stenosis degrees of carotid artery and intracranial arteries, and collateral circulation are evaluated by CDFI and TCCS/TCD.
2. Radiology examination procedures: Before recanalization, enrolled patients receive MRI examinations to determine the presence and the location of cerebral infarction. If necessary, patients receive CT angiography (CTA) , MRI angiography (MRA) or Digital subtraction angiography (DSA) to confirm the degrees of vessel stenosis and occlusion. One week after recanalization, CT and MRI are used to identify the cerebral hemorrhage and newly cerebral infarction.
3. The data collected in this study including:

1) The general information of enrolled subjects, which include age, gender, resident address and telephone number, the history of hypertension, coronary artery diseases, dyslipidemia, diabetes mellitus and smoking.

2. The primary endpoints are: The combination endpoints events of death, cerebral hemorrhage , newly cerebral infarction, hyperperfusion syndrome, residual sternosis≥50% within 30-day after recanalization. The secondary endpoints are the re-current cerebral artery events and the occurence of restenosis during the at least 1 year follow-up period.

4. Statistical analysis plans: The Statistical Package of Social Sciences (SPSS version 22.0) software are used for statistical analysis.

1) Diagnostic test are used to test the sensitivity, specificity and accuracy of ultrasound for evaluating vulnerable plaque by using plaque specimen after CEA as the "gold" standard.

2) The Chi-square test are used to compare the success rate of stenting and CEA. The Cox regression analysis are used to compare the restenosis rate of stenting and CEA.

3) A P<0.05 was considered statistically significance. 5. Quality assurance plan:

1. The medical centers implement the projects are the stroke center awarded by the Stroke Prevention Engineering Committee, the National Health Commission of China. The medical centers have the instruments required in this study.
2. Neurologists, neurosurgeons and vascular ultrasound physicians have received standard training hosted by the Stroke Prevention Engineering Committee, the National Health Commission of China and obtained excellent records.
3. All the centers conduct the project followed the uniform implementation plans and each center guarantee the data input in time and accurately.
4. The project has the unique database and data input in uniform format.
5. There are specific staffs to check the accuracy and completeness of data.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients with carotid artery moderate (50-69%, with symptoms), severe (70-99%, with or without symptoms) stenosis or occlusion diagnosed by CDFI and confirmed by CTA or DSA.

  2) Patient has the indications for carotid artery stenting or CEA according to the guidelines published by the Stroke Prevention Engineering Committee, the National Health Commission of China.

  3) Patient with complete imaging evaluation and can be followed up to at least 1 year.

Exclusion Criteria:

- 1) Patients with non-atherosclerotic carotid artery stenosis or occlusion, such as dissection, aneurysm, arteritis, cardiac embolism and et al.

2) Patients with cerebral hemorrhage. 3) Pregnant

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with carotid artery moderate (50-69%), severe (70-99%) stenosis or occlusion, who needs recanalization by CEA or stenting.
Sampling Method: Non-Probability Sample
Enrollment: 1213 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
The rate of combination endpoints events including death, cerebral hemorrhage , newly cerebral infarction, hyperperfusion syndrome,and residual sternosis≥50%. | within 30-day after recanalization.
  The rate of combination endpoints events, including death, cerebral hemorrhage , newly cerebral infarction, hyperperfusion syndrome, and residual sternosis≥50%

SECONDARY OUTCOMES:
the rate of re-current cerebral artery events and the occurence of restenosis | during the at least 1 year follow-up period
  the rate of re-current cerebral artery events and the occurence of restenosis

CONTACTS AND LOCATIONS:
Overall Officials: Yang Hua, MD, Principal Investigator — No.45 Changchun Road, Beijing,100053, China
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No